CLINICAL TRIAL: NCT02622620
Title: Study on Neuroepithelial Tumor Grading and Pseudoprogression After Glioma Therapy Using Advanced Functional MRI Techniques
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Tang-Du Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2014JZ2-007
Record Dates: First submitted 2015-11-18; First posted 2015-12-04 (Estimated); Last update posted 2016-03-29 (Estimated); Status verified 2016-03

CONDITIONS: Glioma; Neoplasms
Keywords: dynamic contrast-enhanced MR imaging; three-dimensional arterial spin labeling; diffusion-weighted imaging
MeSH Terms: conditions — Glioma; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with glioma: Patients with high-grade glioma (glioblastoma multiforme or anaplastic astrocytoma), who receive concurrent chemoradiation (CCRT) with temozolomide

SUMMARY:
Contrast-enhanced MRI is the most common way for evaluating neuroepithelial tumor grading and monitoring for tumor recurrence,but the ability to predict tumor behavior remains very limited.In this study, the investigators will use multi-b-value diffusion-weighted imaging(DWI),three-dimensional arterial spin labeling(3D-ASL) and dynamic contrast-enhanced MRI imaging(DCE) to evaluate neuroepithelial tumor grading and monitor for tumor recurrence.

DETAILED DESCRIPTION:
Glioma is classified into 4 grades, with worse prognosis for more advanced grades.Previous studies have suggested that different therapeutic strategies should be applied for gliomas at different grades,so glioma grading before the operation is therefore of important clinical significance for guiding the grade-dependent therapeutic strategy.

Combination temozolomide and radiation significantly prolongs survival compared with radiation alone and has become standard treatment for Patients with high-grade glioma. Response assessment in these patients is difficult as a result of the frequent occurrence of early imaging changes indistinguishable from tumor progression, termed pseudoprogression. The majority of patients remain clinically stable. It is often unclear whether current therapy should be maintained or second-line therapy initiated.

The ADC value can potentially reveal the differences in cellularity and nuclear atypia of gliomas1. Theoretically, high cellularity in advanced gliomas may impede free water diffusion and thus lead to a decreased ADC value.In several previous studies,recurrent tumors have shows significantly higher cellularity than those shown by pseudoprogression.Such high cellularity is associated with relative reductions in extracellular space when compared with low cellularity, resulting in decreased diffusivity of water molecules in the former circumstance when compared with the latter. DWI measures the degree of water diffusion within tissue Apparent diffusion coefficient (ADC) values quantify the mobility of water molecules at the cellular level, holding the potential to differentiate between necrosis, edema and recurrent tumor.

A potential mechanism of pseudoprogression is that radiation-induced vascular changes may lead to focal transient increase in gadolinium enhancement.Three-dimensional arterial spin labeling(3D-ASL) and dynamic contrast-enhanced (DCE) MRI imaging provides a noninvasive means for quantifying tumor vascular properties.

ELIGIBILITY:
Inclusion Criteria:

* Among the patients with high-grade glioma (glioblastoma multiforme or anaplastic astrocytoma), who received concurrent chemoradiation (CCRT) with temozolomide, the patients show the measurable enhancing portion (1 cm in the long diameter according to the RANO criteria) in the immediate f/up MRI after CCRT.

Exclusion Criteria:

* Among the patients with high-grade glioma (glioblastoma multiforme or anaplastic astrocytoma), who received concurrent chemoradiation (CCRT) with temozolomide, the patients do not show the measurable enhancing portion (1 cm in the long diameter according to the RANO criteria) in the immediate f/up MRI after CCRT.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with high-grade glioma (glioblastoma multiforme or anaplastic astrocytoma), who receive concurrent chemoradiation (CCRT) with temozolomide
Sampling Method: Probability Sample
Enrollment: 86 (Estimated)
Dates: Start 2016-07; Primary Completion 2018-11 (Estimated); Study Completion 2018-11 (Estimated)

PRIMARY OUTCOMES:
To prospectively acquire multiparameter MR variables at 3T MRI from treated high grade glioma patients to assign tissue signatures for tumor recurrence and pseudoprogression as established by pathologic examination | 24 months

SECONDARY OUTCOMES:
To compare the predictive values of the multiparameter MR tissue signatures acquired at 3T | 24 months

REFERENCES:
- [Derived] Yan LF, Sun YZ, Zhao SS, Hu YC, Han Y, Li G, Zhang X, Tian Q, Liu ZC, Yang Y, Nan HY, Yu Y, Sun Q, Zhang J, Chen P, Hu B, Li F, Han TH, Wang W, Cui GB. Perfusion, Diffusion, Or Brain Tumor Barrier Integrity: Which Represents The Glioma Features Best? Cancer Manag Res. 2019 Nov 27;11:9989-10000. doi: 10.2147/CMAR.S197839. eCollection 2019. PMID 31819632
- [Derived] Liu ZC, Yan LF, Hu YC, Sun YZ, Tian Q, Nan HY, Yu Y, Sun Q, Wang W, Cui GB. Combination of IVIM-DWI and 3D-ASL for differentiating true progression from pseudoprogression of Glioblastoma multiforme after concurrent chemoradiotherapy: study protocol of a prospective diagnostic trial. BMC Med Imaging. 2017 Feb 1;17(1):10. doi: 10.1186/s12880-017-0183-y. PMID 28143434